CLINICAL TRIAL: NCT06515782
Title: Effect of Fasting Mimicking Diet on Measures of Inflammatory Disease in Relapsing Multiple Sclerosis (RMS) Patients Treated With Standard Disease Modifying Therapies
Brief Title: Effect of a Fasting Mimicking Diet on Patients With Multiple Sclerosis (FMDMS)
Acronym: FMDMS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Margaret Burnett, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: HS-21-00212
Record Dates: First submitted 2023-12-04; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Multiple Sclerosis
Keywords: fasting; Mediterranean diet; body composition; quality of life
MeSH Terms: conditions — Multiple Sclerosis; Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: FMD + Mediterranean Diet (Experimental): In the first 6 months, participants will start the Mediterranean diet and undergo 3 cycles of FMD. Participants will then switch to the Mediterranean diet alone for another 6 months.
  Interventions: Other: Med Diet. Investigators would like to see what differences a Mediterranean Diet makes to the status of patients with Multiple Sclerosis.
- Arm 2: Mediterranean Diet + FMD (Active Comparator): Participants will start with Mediterranean diet alone for the first 6 months and after that they will undergo FMD for 3 cycles while still on a Mediterranean diet.
  Interventions: Other: Med Diet. Investigators would like to see what differences a Mediterranean Diet makes to the status of patients with Multiple Sclerosis.

INTERVENTIONS:
Other: Med Diet. Investigators would like to see what differences a Mediterranean Diet makes to the status of patients with Multiple Sclerosis. — In one group investigators will look at the Med diet alone for 6 months. Then investigators will have the patients add on 3 rounds of FMD.
  In the other group, patients will do Med diet and FMD for 6 months followed by Med diet alone for 6 months. This will allow investigators to look for a diminution in effect of the Med diet 6 months after the last FMD.
  Other Names: Is there an additional change to status when patients undergo 3 rounds of fast mimicking diet?

SUMMARY:
In the proposed study, investigators will assess the safety and feasibility of cycles of a fasting mimicking diet (FMD) and its effect on Multiple Sclerosis Quality of Life (MSQOL) in relapsing MS (RMS) patients treated with standard disease modifying therapies (FMDMS).

To test the primary hypothesis, investigators will compare the composite quality of life score in terms of improvement in disability, fatigue, and cognitive function with the fasting protocol, as compared to a Mediterranean diet (control) group alone. Further, investigators hypothesize that the effects will remain for at least 6-months after the last FMD cycle. The Mediterranean diet (MD) has been chosen as the control diet to minimize baseline dietary differences among patients. It has been trialed for feasibility in Multiple Sclerosis patients and used in a previous human FMD trial for MS patients where a FMD followed by MD was shown to have positive effects on people with MS.

DETAILED DESCRIPTION:
The study design is a cross-over randomized, controlled trial that includes two arms in which all patients will be on a MD for twelve months. One group will be on MD alone for 6 months and then do 3 rounds of a standardized 7-day FMD dietary regimen every 2 months. The other group will do the 3 cycles of FMD during the first 6 months, and the subsequent 6 months on the MD alone. This will allow investigators to test FMD effects on a defined background diet as well as tease out the effects of that diet alone. In addition, investigators will be able to assess long term effects of a FMD on an autoimmune disease.

Preliminary data from a phase I clinical study in MS suggest that a FMD is safe, feasible, and potentially effective in relapsing-remitting multiple sclerosis (RRMS) patients (registered in Clinical Trials ID: NCT01538355). This study demonstrated a positive effect on health-related quality of life (HRQOL) components and a small effect on disability after one round FMD followed by a Mediterranean diet for 5 months.

A successful trial will provide relevant information about the efficacy and safety of these dietary interventions in MS patients and help confirm the positive effects seen in previous studies. In addition it is designed to elucidate the physiologic and immunologic effects of dietary changes and could help clarify the complex interactions between nutrition and autoimmune disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS (AJ Thompson et al 2018)
* Able to give informed consent
* Able to tolerate MRI
* Age 18 to 55 years
* Disease duration 6 months to 20 years (included)
* EDSS 0 to 6
* No change in immunomodulatory therapy in the 6 months prior to enrollment (not on immunomodulatory therapy is acceptable)
* No glucocorticoid use within 30 days prior to screening
* No serologic evidence of vitamin B12 deficiency or hypothyroidism
* No Vitamin D deficiency (< 30 ng/ml)

Exclusion Criteria:

* Relapse < 60 days.
* Any active or chronic infection (e.g. HIV, Syphilis, untreated TB)
* Previous history of a malignancy other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
* Severely limited life expectancy by another co-morbid illness
* History of previous diagnosis of myelodysplasia or previous hematologic disease or current clinically relevant abnormalities of white blood cell counts
* Pregnancy or risk of pregnancy (this includes patients who are unwilling to practice active contraception during the duration of the study)
* eGFR < 60 mL/min/1.73m2 or known renal failure or inability to undergo MRI examination
* Inability to give written informed consent in accordance with research ethics board guidelines
* Known alimentary allergy or intolerance to any of the ingredients of the FMD regimen or the presence of diabetes
* Underweight

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Health-related Quality of Life (HRQOL) | 12 months
  Improvement in disability, fatigue and cognitive function. Scale and composite scores range from 0 to 100, where a higher score indicates a better QOL.

SECONDARY OUTCOMES:
Assessing Safety and Tolerability of a FMD in MS: Compliance and Serious Adverse Events | 12 months
  To evaluate the safety and tolerability of a FMD will be assessed using assessed using a standardized safety questionnaire. Adverse events will be scored utilizing Common Terminology Criteria for Adverse Events (CTCAE)
To evaluate the effect on clinical measures of neurological status: Annualized relapse rate | 12 months
  Relapses will be verified by clinical visit, history, and possible imaging. Rates will be analyzed per year
To evaluate the effect on clinical measures of neurological status: EDSS | 12 months
  Expanded disability status score (EDSS): A verified instrument to verify the disability of the patient. The score range from 0-10 with larger numbers indicating worse disability.
To evaluate the effect on clinical measures of neurological status: depression, anxiety | 12 months
  We will assess anxiety and depression using Hospital Anxiety and Depression Scale (HADS). The score range from 0-21 with smaller numbers being better
To evaluate body composition | 12 months
  Changes in body composition: BMI (Weight and height will be combined to report BMI: kg/m^2)
To evaluate IGF-1 changes | 12 months
  Changes in Insulin like growth factor 1 (IGF-1) (ng/mL) which measure FMD effectiveness and a lower animal protein intake.
To estimate changes in measures of disease activity in the central nervous system (CNS) | 12 months
  Number and volume of new and enlarging lesions detected by MRI. Units Cm^2
To estimate changes in measures of disease activity in the central nervous system (CNS) | 12 months
  Changes in serum concentrations of neurofilament light chain (NF-L). Units: ng/L
To evaluate alterations in immune function by assessing changes in cell counts, serum cytokines and secretion patterns, with a focus on pro-inflammatory cytokines IL-2, interferon-gamma (IFNγ), and IL-17A, and the regulatory cytokine, IL-10. Units: pg/mL | 12 months
  It is known that lymphocyte counts decrease during fasting.
To evaluate changes following the FMD in the composition and function of the gut microbiota which influences immune function in the T and B cells compartment in the blood. | 12 months
  It has been shown that patients with MS have moderate alterations of gut microbial communities. Units: μm

CONTACTS AND LOCATIONS:
Overall Officials: Margaret E Burnett, MD, Principal Investigator — University of Southern California Keck School of Medicine
Locations (1):
- Keck School of Medicine of the University of Southern California, Los Angeles, California, United States